CLINICAL TRIAL: NCT03984188
Title: Effectiveness of Low-Dose Theophylline for the Management of Biomass-Associated COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Trishul Siddharthan, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20201523; 1K23HL146946-01 (NIH); IRB00209008 (Other: Johns Hopkins University)
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: COPD; COPD Exacerbation; COPD Exacerbation Acute; Pollution Related Respiratory Disorder; Pollution; Exposure
Keywords: Biomass Associated COPD; Low-dose Theophylline
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose Theophylline Group (Experimental): Participant in this group will receive low-dose theophylline in addition to standard care, per World Health Organization (WHO) guidelines for management of Chronic Obstructive Pulmonary Disease (COPD) treatment, over a one year period.
  Interventions: Drug: Theophylline ER; Other: Standard of Care Treatment
- Placebo Group (Placebo Comparator): Participant in this group will receive a placebo in addition to standard care, per World Health Organization (WHO) guidelines for management of Chronic Obstructive Pulmonary Disease (COPD) treatment.
  Interventions: Drug: Placebo oral tablet; Other: Standard of Care Treatment

INTERVENTIONS:
Drug: Theophylline ER — 200 mg extended release (ER) low-dose theophylline taken orally daily
  Other Names: Low-dose Theophylline
  Arms: Low-dose Theophylline Group
Drug: Placebo oral tablet — Manufactured methylcellulose placebo tablet taken orally daily
  Arms: Placebo Group
Other: Standard of Care Treatment — Per World Health Organization (WHO) guidelines for management of Chronic Obstructive Pulmonary Disease (COPD) treatment

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death worldwide, and over 90% of COPD-related deaths occurring in low- and middle-income countries (LMICs). Household air pollution (HAP) - from burning solid fuels such as wood, dung, agricultural crop waste, and coal for energy - is the primary risk factor for COPD in these settings. Biomass-related COPD has a distinct histopathology, phenotype and inflammatory profile when compared to tobacco mediated COPD. Despite the high global burden of biomass-related disease, little is known about the effectiveness of pharmacotherapies for biomass-related COPD; to date, no clinical trials have focused specifically on treatment of biomass-related COPD. This study proposes to assess the health impact of biomass-related COPD and test the effectiveness of low dose theophylline compared to standard therapy among adults with biomass-related COPD in Uganda with the aim to assess whether low-dose theophylline improves respiratory symptoms, decreases the inflammatory profile of serum biomarkers and whether administration attenuates the effect of HAP on lung function. The study additionally aims to assess whether low-dose theophylline is a cost-effective intervention based on the incremental cost-effectiveness ratio and a range of willingness to pay thresholds.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Full-time resident of study area
3. Post-bronchodilator FEV1/FVC < the lower limit of normal of the Global Lung Initiative Mixed Ethnic reference population
4. Grade B-D COPD
5. Daily biomass exposure

Exclusion Criteria:

1. Plans to move within one year
2. Uncontrolled hypertension
3. Pregnancy (assessed by urine pregnancy test among women of childbearing age/menstrual history)
4. Current use of chronic respiratory medications (Long acting Beta 2 Antagonists (LABA), Long-acting muscarinic antagonist (LAMA), inhaled corticosteroid (ICS))
5. History of post-treatment pulmonary tuberculosis
6. ≥10 pack year tobacco smoking history
7. Known intolerance or contraindication to theophylline.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trishul Siddharthan, MD, Principal Investigator — University of Miami
Locations (2):
- Uganda (2):
  - Makerere Lung Institute, Kampala
  - Nakaseke Hospital, Nakaseke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonjour S, Adair-Rohani H, Wolf J, Bruce NG, Mehta S, Pruss-Ustun A, Lahiff M, Rehfuess EA, Mishra V, Smith KR. Solid fuel use for household cooking: country and regional estimates for 1980-2010. Environ Health Perspect. 2013 Jul;121(7):784-90. doi: 10.1289/ehp.1205987. Epub 2013 May 3. PMID 23674502
- [Background] Siddharthan T, Grigsby MR, Goodman D, Chowdhury M, Rubinstein A, Irazola V, Gutierrez L, Miranda JJ, Bernabe-Ortiz A, Alam D, Kirenga B, Jones R, van Gemert F, Wise RA, Checkley W. Association between Household Air Pollution Exposure and Chronic Obstructive Pulmonary Disease Outcomes in 13 Low- and Middle-Income Country Settings. Am J Respir Crit Care Med. 2018 Mar 1;197(5):611-620. doi: 10.1164/rccm.201709-1861OC. PMID 29323928
- [Background] Moran-Mendoza O, Perez-Padilla JR, Salazar-Flores M, Vazquez-Alfaro F. Wood smoke-associated lung disease: a clinical, functional, radiological and pathological description. Int J Tuberc Lung Dis. 2008 Sep;12(9):1092-8. PMID 18713510
- [Background] Perez-Padilla R, Ramirez-Venegas A, Sansores-Martinez R. Clinical Characteristics of Patients With Biomass Smoke-Associated COPD and Chronic Bronchitis, 2004-2014. Chronic Obstr Pulm Dis. 2014 May 6;1(1):23-32. doi: 10.15326/jcopdf.1.1.2013.0004. PMID 28848808
- [Background] Ait-Khaled N, Enarson D, Bousquet J. Chronic respiratory diseases in developing countries: the burden and strategies for prevention and management. Bull World Health Organ. 2001;79(10):971-9. Epub 2001 Nov 1. PMID 11693980
- [Background] Beran D, Zar HJ, Perrin C, Menezes AM, Burney P; Forum of International Respiratory Societies working group collaboration. Burden of asthma and chronic obstructive pulmonary disease and access to essential medicines in low-income and middle-income countries. Lancet Respir Med. 2015 Feb;3(2):159-170. doi: 10.1016/S2213-2600(15)00004-1. PMID 25680912
- [Background] Barnes PJ. Theophylline in chronic obstructive pulmonary disease: new horizons. Proc Am Thorac Soc. 2005;2(4):334-9; discussion 340-1. doi: 10.1513/pats.200504-024SR. PMID 16267358
- [Background] Ford PA, Durham AL, Russell RE, Gordon F, Adcock IM, Barnes PJ. Treatment effects of low-dose theophylline combined with an inhaled corticosteroid in COPD. Chest. 2010 Jun;137(6):1338-44. doi: 10.1378/chest.09-2363. Epub 2010 Mar 18. PMID 20299628
- [Background] Rivera RM, Cosio MG, Ghezzo H, Salazar M, Perez-Padilla R. Comparison of lung morphology in COPD secondary to cigarette and biomass smoke. Int J Tuberc Lung Dis. 2008 Aug;12(8):972-7. PMID 18647460
- [Background] Mendis S, Fukino K, Cameron A, Laing R, Filipe A Jr, Khatib O, Leowski J, Ewen M. The availability and affordability of selected essential medicines for chronic diseases in six low- and middle-income countries. Bull World Health Organ. 2007 Apr;85(4):279-88. doi: 10.2471/blt.06.033647. PMID 17546309
- [Background] Zhou Y, Wang X, Zeng X, Qiu R, Xie J, Liu S, Zheng J, Zhong N, Ran P. Positive benefits of theophylline in a randomized, double-blind, parallel-group, placebo-controlled study of low-dose, slow-release theophylline in the treatment of COPD for 1 year. Respirology. 2006 Sep;11(5):603-10. doi: 10.1111/j.1440-1843.2006.00897.x. PMID 16916334
- [Derived] Siddharthan T, Pollard SL, Jackson P, Robertson NM, Wosu AC, Rahman N, Padalkar R, Sekitoleko I, Namazzi E, Alupo P, Hurst JR, Kalyesubula R, Dowdy D, Wise R, Barnes PJ, Checkley W, Kirenga B. Effectiveness of low-dose theophylline for the management of biomass-associated COPD (LODOT-BCOPD): study protocol for a randomized controlled trial. Trials. 2021 Mar 16;22(1):213. doi: 10.1186/s13063-021-05163-2. PMID 33726828

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is a discrepancy between the protocol section enrollment number vs the participants that started in the participant flow due to one participant decided not to proceed in the study after they consented and were enrolled but left the study just prior to randomization and therefore did not proceed in the study.
Period: Overall Study
Arm/Group | Low-dose Theophylline Group | Placebo Group
Started | 50 | 49
6 Months | 42 | 47
Completed | 39 | 41
Not Completed | 11 | 8
Not completed — Death | 2 | 4
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Theophylline Group | Placebo Group | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 19 | 19 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 20 | 24 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 49 | 99
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in St. George Respiratory Questionnaire (SGRQ) Scores
Description: The SGRQ comprises of 50 items and consists of two parts. The first part pertains to symptoms and the second pertains to functional status as well as social and psychological impact of disease. Overall scores ranges between 0 and 100 with higher scores indicating more limitations.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-dose Theophylline Group | Placebo Group
Number analyzed (Participants) | 39 | 41
score on a scale | 39.02 (21.00) | 45.06 (16.87)

2. Secondary Outcome: Change in Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 measures how much air a person can exhale during a forced breath. The amount of air exhaled during the first second measured in liters.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Low-dose Theophylline Group | Placebo Group
Number analyzed (Participants) | 38 | 38
Liters | 1.40 (0.51) | 1.45 (0.58)

3. Secondary Outcome: Change in Forced Vital Capacity (FVC)
Description: FVC measures how much air a person can exhale at the end of a forced breath measured in liters.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Low-dose Theophylline Group | Placebo Group
Number analyzed (Participants) | 38 | 38
Liters | 2.47 (0.68) | 2.58 (0.81)

4. Secondary Outcome: Change in Forced Vital Capacity (FVC)
Description: FVC measures how much air a person can exhale at the end of a forced breath measured in liters.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Low-dose Theophylline Group | Placebo Group
Number analyzed (Participants) | 42 | 44
Liters | 2.51 (0.68) | 2.52 (0.84)

5. Secondary Outcome: Change in St. George Respiratory Questionnaire (SGRQ) Scores
Description: as for outcome 1
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-dose Theophylline Group | Placebo Group
Number analyzed (Participants) | 42 | 47
score on a scale | 37.86 (21.37) | 44.45 (19.48)

6. Secondary Outcome: Change in Forced Expiratory Volume in One Second (FEV1)
Description: as for outcome 2
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Low-dose Theophylline Group | Placebo Group
Number analyzed (Participants) | 42 | 44
Liters | 1.40 (0.51) | 1.40 (0.62)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Low-dose Theophylline Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 2/50 | 4/49
Serious Adverse Events (participants affected / at risk) | 5/50 | 3/49
Other Adverse Events (participants affected / at risk) | 26/50 | 19/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Theophylline Group (N=50) | Placebo Group (N=49)
Hospitalization for Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hospitalization for Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalization for anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalization for failure to thrive (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-dose Theophylline Group (N=50) | Placebo Group (N=49)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Arthalgia/Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Change in urinary frequency (Renal and urinary disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03984188/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03984188/SAP_001.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03984188/ICF_002.pdf